CLINICAL TRIAL: NCT03316989
Title: Melatonin Levels and Obesity
Brief Title: Melatonin Levels and the Relation to Obesity and the Metabolic Syndrome in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Orit Hamiel, Head department of Pediatric Endocrinology, Sheba Medical Center
Other Study IDs: SHEBA-09-7461-OH-CTIL
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Metabolic Syndrome Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- obese children: Children and adolescents with BMI according to the CDC greater that 95%ile
- normal weight: Children and adolescents with BMI according to the CDC less than the 85%ile
- obese with the MetS: obese children with metabolic syndrome compared to obese children with out the MetS and normal weight children

SUMMARY:
Background: Melatonin is a neurohormone that regulates the circadian rhythm by translating photoperiodic information from the eyes to the brain.

Working hypothesis and aims: There is a possible link between circadian rhythm regulation and glucose homeostasis through melatonin pathways. We aim to examine the relation between melatonin levels and degree of obesity , in children and adolescents in different pubertal stages.

Methods: The study group will include 24 children and adolescents in various stages of pubertal development. Participants will be categorized into 3 groups: 1) normal-weight, 2) obese subjects with metabolic syndrome, 3) obese without metabolic syndrome. Melatonin levels will be measured using saliva during the night.

Expected results: We expect to find a relation between melatonin levels to the metrics of metabolic syndrome, sleep duration, number of television viewing hours and sense of depression.

Importance: Childhood obesity is recognized as a major medical and public health problem and is strongly associated with many serious medical complications including the metabolic syndrome and Type 2 diabetes (T2DM). It is important to understand mechanisms involved in the development of obesity and hyperinsulinemia.

Probable implications to Medicine: Foreseeing a connection between melatonin levels and the degree of obesity and metabolic syndrome in children and adolescents, we would recommend addressing duration of sleep while treating obesity.

DETAILED DESCRIPTION:
Background: Melatonin is a neurohormone that regulates the circadian rhythm by translating photoperiodic information from the eyes to the brain. MTNR1B , is one of melatonin receptors which is expressed in the retina, in the brain and in pancreatic tissue. In Genome Wide Association studies a SNP in the intronic variant in MTNR1B was found to be to in association with elevated fasting plasma glucose and with increased risk of T2DM among lean and obese adults and children.

Working hypothesis and aims: There is a possible link between circadian rhythm regulation and glucose homeostasis through melatonin pathways. We aim to examine the relation between melatonin levels and degree of obesity and the metabolic syndrome, in children and adolescents in different pubertal stages.

Methods: The study group will include twenty-four children and adolescents in various stages of pubertal development. Participants will be categorized into three groups: 1) normal-weight, 2) obese subjects with metabolic syndrome, 3) obese without metabolic syndrome. Melatonin levels will be measured using saliva during the night. Each child will be measured for height, weight, waist circumference and blood pressure. Fasting insulin, glucose and lipid profile will be taken. Each child will fill out questionnaires about depression, sleep quality and television usage.

Expected results: We expect to find a relation between melatonin levels to the metrics of metabolic syndrome, sleep duration, number of television viewing hours and sense of depression. We expect to find lower levels of melatonin in the group of obese children with metabolic syndrome during night time. We expect that children with lower levels of melatonin should report on fewer hours of sleep, more hours of watching television and feeling more depressed.

Importance: Childhood obesity is recognized as a major medical and public health problem and is strongly associated with many serious medical complications including the metabolic syndrome and Type 2 diabetes (T2DM). It is important to understand mechanisms involved in the development of obesity and hyperinsulinemia.

Probable implications to Medicine: Foreseeing a connection between melatonin levels and the degree of obesity and metabolic syndrome in children and adolescents, we would recommend addressing duration of sleep while treating obesity.

ELIGIBILITY:
Inclusion Criteria:

* obese children
* normal weight children

Exclusion Criteria:

* genetic diseases
* medication that may affect melatonin secretion
* sleep inducing medication

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children and adolescents with obesity and normal weight
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-06-29 (Actual); Primary Completion 2013-05-30 (Actual); Study Completion 2013-05-30 (Actual)

PRIMARY OUTCOMES:
Melatonin levels | 8 hours
  Melatonin levels in the saliva during the evening and night